CLINICAL TRIAL: NCT05996640
Title: Investigating Patient Preferences and Experiences of Waiting for Elective Heart Surgery: a Cross-sectional Online Survey
Brief Title: Patient Preferences and Experiences of Waiting for Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 319498
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is study does not use an intervention — This is study does not use an intervention. A survey will be used to collected data on patients' experiences and preferences about waiting list for heart surgery.

SUMMARY:
Waiting for heart surgery could be difficult and anxiety-provoking for some patients. Research suggests that some specific factors (e.g., individual coping strategies, communication with the clinical team, having a more active role in care decision-making) could reduce the stress associated with waiting. However, most of this research has looked at patients waiting for other types of surgery (e.g., cancer surgery). Therefore, more research focusing on patients waiting for heart surgery is needed.

This project aims to investigate patients' experiences, perceptions and preferences about waiting for elective (non-emergency) heart surgery across four London-based National Health Service (NHS) hospitals that belong to King's Health Partners (KHP): Royal Brompton, Harefield, St Thomas', and King's College hospitals. The project is led by the research team at King's Improvement Science, (King's College London), in collaboration with clinicians and patients with lived experience of waiting for heart surgery.

This project will look at:

* how patients feel their heart condition affects their day-to-day life;
* how patients experience being on a waiting list;
* what factors patients consider as most important for their upcoming surgery (e.g. to have their surgery as soon as possible, at their nearest hospital, or carried out by a specific surgeon);
* patients' opinions about how the heart surgery waiting list process could be improved.

Adult patients (>18 years old) waiting for elective heart surgery at the four hospitals listed above will be invited, via a text message and a letter, to complete an online survey (i.e. a list of questions). Completing reading study information and completing the survey will likely take approximately 30 minutes. The survey will be open for 8 weeks in total.

Findings from this project, together with other work looking at clinical processes and outcomes across heart surgery services at the four KHP hospitals, will inform a wider quality improvement project.

ELIGIBILITY:
Inclusion Criteria:

* being on a waiting list for elective cardiac surgery under any of the following surgical prioritisation categories P2, P3, and P4;
* being at least 18 years old;
* being on a waiting list for cardiac surgery across any of the four KHP participating sites: RBH, HH, STH, and KCH.

Exclusion Criteria:

* being on a waiting list for cardiac surgery at sites other than Royal Brompton Hospital, Harefield Hospital, St Thomas Hospital, and King's College Hospital;
* not having any recorded contact details in the form of mobile phone and home address

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the NHS guide for surgical prioritisation, waiting lists for elective surgery are grouped into four priority categories: P1 includes emergency patients (requiring surgery within 24 hours, therefore they are not on elective cardiac surgery waiting lists); P2 includes patients who require surgery within 4 weeks; P3 and P4 are patients who require surgery within 3 months, and between 3-6 months, respectively.
  The population of interest in this study is composed by patients in the P2, P3 and P4 categories whose most common diagnoses are coronary heart disease, aortic stenosis, mitral regurgitation, and aortic aneurysm. Accordingly, the most commonly performed surgeries within the above categories are coronary artery bypass grafts (CABGs), aortic valve replacement, mitral valve repair or replacement and aortic aneurysm repair.
Sampling Method: Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2023-08-14 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Patient experience | 8 weeks
  ratings on impact of heart condition on life
Patient preferences | 8 weeks
  qualitative description of preferences about service improvement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russo M, Richards KL, Kumar R, Burridge J, Chaplin H, Chua KC, Hardy D, Avlonitis VS, Baig K, Bhudia S, Noorani A, Khan H, Petrou M. Patient experience and preference while waiting for elective cardiac surgery: a mixed-methods cross-sectional survey across four major National Health Service hospitals in London. BMJ Open. 2026 Jan 21;16(1):e102185. doi: 10.1136/bmjopen-2025-102185. PMID 41565334
- [Derived] Russo M, Watson K, Richards K, Olive RR, Krausova B, Kumar R, Burridge J, Goulding L, Chua KC, Hardy D, Vassilios A, Kamran B, Bhudia S, Alia N, Habib K, Sevdalis N, Petrou M. Study protocol for a cross-sectional online survey investigating patient preferences and experiences of waiting for elective cardiac surgery. BMJ Open. 2024 Mar 4;14(3):e079692. doi: 10.1136/bmjopen-2023-079692. PMID 38443077